CLINICAL TRIAL: NCT01880203
Title: Diagnostic Value of Molecular Cytological Analysis (CMA) and Shear Wave Elastography ShearWave (SWE) in Patients With a Thyroid Nodule With Indeterminate Cytology: Feasibility Study
Acronym: SWEETMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Fondation avenir (Unknown); laboratoire Genzyme (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SWEETMAC
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Thyroid Node; Indeterminate Cytology; Surgery Indication
Keywords: thyroid; elastography SWE; indeterminate cytology
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- aspiration for Molecular Cytogenetic Analysis. (Experimental)
  Interventions: Procedure: aspiration in thyroid node for Molecular Cytogenetic Analysis.

INTERVENTIONS:
Procedure: aspiration in thyroid node for Molecular Cytogenetic Analysis.
  Other Names: cervical ultrasound with elastography SWE followed by a new ultrasound-guided fine needle aspiration for Molecular Cytogenetic Analysis.

SUMMARY:
The purpose of the study is to investigate the contribution of molecular cytological analysis (CMA) and shear wave elastography ShearWave (SWE) in the diagnosis of nodules with indeterminate cytology (IC)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with thyroid nodules ≥ 15 mm with an indeterminate cytology (IC) older than 6 months, for which a surgical indication was raised

  * vesicular lesion of undetermined significance
  * follicular neoplasm or Hurthle cells
  * lesion suspicious for malignancy
* Confirmation of indeterminate cytology (IC) replay centralized
* Patient affiliated to a social security scheme
* Informed consent and signed

Exclusion Criteria:

* Thyroid node <15 mm
* Nodules coalescing preventing proper individualization of targeted nodule
* Indeterminate cytology older than six months
* Nodules with indeterminate cytology not, ie non-diagnostic cytology, benign and malignant cytology cytology
* Major subject to a measure of legal protection or unable to consent
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic performance of the AMC and SWE elastography | at inclusion, before surgery
  Evaluate the diagnostic performance of the AMC and SWE elastography in patients with a thyroid nodule CI taking as reference the histology of the nodule.

SECONDARY OUTCOMES:
evaluate the diagnostic performance of elastography SWE | at inclusion, before surgery
  For elastography SWE validate decision thresholds for the parameters of elasticity of thyroid nodules, and evaluate the diagnostic performance of elastography SWE combined with those of the standard ultrasound.
Establish a combined diagnostic score results of elastography | at inclusion, before surgery
  Establish a combined diagnostic score results of elastography, the standard ultrasound and molecular analysis

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre François BACLESSE, Caen, Calvados
  - CHU, Caen, Calvados
  - Hôpital Américain de Paris, Neuilly-sur-Seine
  - Hôpital Pitié-salpétrière, Paris

REFERENCES:
- [Derived] Bardet S, Goardon N, Lequesne J, Vaur D, Ciappuccini R, Leconte A, Monpeyssen H, Saguet-Rysanek V, Clarisse B, Lasne-Cardon A, Menegaux F, Leenhardt L, Buffet C. Diagnostic and prognostic value of a 7-panel mutation testing in thyroid nodules with indeterminate cytology: the SWEETMAC study. Endocrine. 2021 Feb;71(2):407-417. doi: 10.1007/s12020-020-02411-4. Epub 2020 Jul 7. PMID 32638211